CLINICAL TRIAL: NCT00889954
Title: Administration of Her2 Chimeric Receptor and TGFbeta Dominant Negative Receptor (DNR) Expressing EBV Specific Lymphocytes for Subjects With Advanced Her2 Positive Malignancy (HERCREEM)
Brief Title: Her2 and TGFBeta Cytotoxic T Cells in Treatment of Her2 Positive Malignancy
Acronym: HERCREEM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Stephen Gottschalk, Associate Professor Pediatric Hematology/Oncology Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24486-HERCREEM; HERCREEM (Other: Baylor College of Medicine)
Record Dates: First submitted 2009-04-24; First posted 2009-04-29 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: HER2 Positive Malignancies
Keywords: EBV+; Her2; TGFBeta; EBV positive; HER 2 positive malignancy; cytotoxic T lymphocytes
MeSH Terms: conditions — Camurati-Engelmann Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TGFBeta resistant HER2/EBV-CTLs (Experimental): The following dose levels will be evaluated:
  Dose Level 1: 1 x 10^4 cells/m^2
  Dose Level 2: 3 x 10^4 cells/m^2
  Dose Level 5: 1 x 10^6 cells/m^2
  Dose Level 6: 3 x 10^6 cells/m^2
  Dose Level 7: 1 x 10^7 cells/m^2
  Dose Level 8: 3 x 10^7 cells/m^2
  Dose Level 9:1 x 10^8 cells/m^2
  Interventions: Biological: TGFBeta resistant HER2/EBV-CTLs

INTERVENTIONS:
Biological: TGFBeta resistant HER2/EBV-CTLs — Each patient will receive one injection of the TGFBeta resistant HER2/EBV-specific CTLs. Each pt will be followed for 6 weeks after the CTL infusion for evaluation of dose limiting toxicity (DLT).
  Patients may receive up to six additional doses of the T cells at 6 to 12 weeks intervals.
  Other Names: HER2-DNR EBV T cells

SUMMARY:
Patients have advanced stage cancer. This study is a gene transfer research study using special immune cells.

The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Investigators hope that both will work better together. Antibodies are proteins that protect the body from diseases caused from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting blood cells that can kill other cells, including tumor cells or cells that are infected with germs. Both antibodies and T cells have been used to treat patients with cancers: they both have shown promise, but have not been strong enough to cure most patients.

T lymphocytes can kill tumor cells but there are normally not enough of them or they are not able to kill all the tumor cells. We have done research in which we have grown "extra" T lymphocytes. We have added genes to those T lymphocytes to help them to recognize tumor cells. Although the results have been promising, we are still doing more research in this area.

Antibodies usually circulate in blood and are secreted by other cells of the immune system in response to the presence of germs or abnormal cells in the body. The antibody used in this study is called anti-HER2 (Human Epidermal Growth Factor Receptor 2). This antibody sticks to HER2-positive cancer cells because of a substance on the outside of these cells called HER2.

DETAILED DESCRIPTION:
The patient will give blood to grow T cells on either one to two separate occasions. Then, the EBV-specific T cells will be made. These cells will be grown and frozen. To get the HER2 antibody (and the CD28) and the DNR to attach to the surface of the EBV-T cells, the antibody gene and the DNR gene will be inserted into the EBV-T cell. This is done with two viruses called retroviruses that have been made for this study. One will carry the antibody gene into the T cell and the other the DNR gene.

When the patient is enrolled on the study, they will be assigned to a dose of HER2-DNR EBV-T cells. The subject will be given one dose of cells into the vein through an IV line. The injection will take between 1 and 10 minutes. The patient will be followed in the clinic after the injection for 1 to 4 hours. The treatment will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

ELIGIBILITY:
INCLUSION CRITERIA:

The patient must meet the following eligibility inclusion criteria at the time of PROCUREMENT:

1. Diagnosis of advanced stage* or metastatic HER2-positive cancer (Immunohistochemistry or reverse transcription-polymerase chain reaction (RT-PCR) is used to determine HER2 positivity)

   Definitions of Malignancies and Advanced Stages:

   Breast ≥Stage IIIb Colon cancer ≥Stage IIIb Esophageal cancer ≥Stage IIIb Gastric carcinoma ≥Stage IIIb Head and Neck cancer Stage IV Lung cancer ≥Stage IIIb Pancreatic cancer Stage IV Prostate cancer Stage IV

   *it is expected that the majority of patients who will be accrued on the protocol will have one of the HER2-positive malignancies listed in the table. If the patient's malignancy is not listed we will use ≥ Stage IIIb as the definition of advanced stage disease. If Stage IIIb is not part of the staging system for the individual tumor, Stage IV will be used.

   For World Health Organization grade III and IV brain tumors):patients will be eligible, who have recurrent or progressive disease after front line therapy.
2. Karnofsky/Lansky score of 50 or more
3. EBV seropositive
4. Greater than or equal to 3 years old
5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

The patient must meet the following eligibility criteria to be included for TREATMENT:

1. Diagnosis of advanced stage* or metastatic HER2-positive cancer with disease progressed after receiving at least one prior systemic therapy. (Immunohistochemistry or RT-PCR is used to determine HER2 positivity) *for definition refer to Table above.
2. Greater than or equal to 3 years old.
3. EBV-seropositive
4. Recovered from the acute toxic effects of all prior chemotherapy at least a week before entering this study.
5. Normal echocardiogram (Left ventricular ejection fraction (LVEF) has to be with in normal, institutional limits)

5. Life expectancy 6 weeks or more

7. Karnofsky/Lansky score of 50 or more

8. Bilirubin 3x or less, Aspartate aminotransferase (AST) 5x or less, Serum creatinine 2x or less upper limit of normal, Hgb 9.0 g/dl or more, white blood cells greater than 2,000/ul, absolute neutrophil count greater than 1,000/ul, Platelets greater than 100,000/ul

9. Pulse oximetry 90% or more on room air

10. Sexually active patients must be willing to utilize one of the more effective birth control methods for 6 months after the CTL infusion. Male partner should use a condom. Acceptable forms of birth control include: * oral contraceptives ("the pill"), * intrauterine devices (IUDs), * contraceptive implants under the skin, or contraceptive injections, * condoms with foam.

11. Available autologous transduced EBV-specific cytotoxic T lymphocytes with 15% or more expression of HER2 CAR determined by flow-cytometry and killing of Her2-positive targets 20% or more in cytotoxicity assay.

12. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

Note: Patients must also not receive antineoplastic drugs while on this study since they would kill the infused T cells.

EXCLUSION CRITERIA:

At time of Procurement:

1. Known HIV positivity

At time of Treatment:

1. Severe intercurrent infection
2. Known HIV positivity
3. Pregnant or lactating
4. History of hypersensitivity reactions to murine protein-containing products

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-05; Primary Completion 2015-07 (Actual); Study Completion 2018-01-21 (Actual)

PRIMARY OUTCOMES:
Number of Patients with dose limiting toxicity. | 6 weeks
  Determine safety of one IV injection of autologous TGFBeta-resistant cytotoxic T cells (CTL) directed to Epstein Barr virus (EBV) through their native receptor and HER2 through their chimeric antigen receptor (CAR) in patients with advanced HER2- positive cancers.

SECONDARY OUTCOMES:
Area under the growth curves (AUC) over time for T cell frequencies. | 15 years
  To compare the survival and the immune function of the TGFBeta-resistant and non resistant components of the infused CAR-CTL.
Decrease in tumor after the CTL infusion | 15 years
  To assess the anti-tumor effects of the infused CAR-CTL.

CONTACTS AND LOCATIONS:
Overall Officials: Stepehen Gottschalk, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas